CLINICAL TRIAL: NCT00639314
Title: Randomized Controlled Trial on the Evaluation of Pylorus-ring in Pancreaticoduodenectomy
Brief Title: Trial on the Evaluation of Pylorus-ring in Pancreaticoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wakayama Medical University (Other)
Responsible Party: Second Department of Surgery, Wakayama Medical University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WP-0502
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2010-01

CONDITIONS: Pancreatic Cancer; Bile Duct Cancer; Ampullary Cancer; Duodenal Cancer; Pancreatitis
Keywords: pylorus-preserving pancreaticoduodenectomy; pylorus-resecting pancreaticoduodenectomy; randomized controlled trial; delayed gastric empty; quality of life
MeSH Terms: conditions — Pancreatic Neoplasms; Bile Duct Neoplasms; Duodenal Neoplasms; Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): In PpPD, the proximal duodenum was divided 3-4cm distal to the pylorus ring
  Interventions: Procedure: pylorus-preserving pancreaticoduodenectomy
- 2 (Active Comparator): In PrPD, the stomach is divided just above the pylorus ring. the nearly total stomach more than 95% was preserved.
  Interventions: Procedure: pylorus-resecting pancreaticoduodenectomy

INTERVENTIONS:
Procedure: pylorus-preserving pancreaticoduodenectomy — pylorus-preserving resection is division of the duodenum 3-4cm distal to the pylorus
  Arms: 1
Procedure: pylorus-resecting pancreaticoduodenectomy — In PrPD, the stomach is divided just above the pylorus ring. The nearly total stomach more than 95% was preserved.
  Arms: 2

SUMMARY:
The purpose of this study is to clarify whether resecting pylorus-ring decreases delayed gastric emptying after pancreaticoduodenectomy and improves postoperative quality of life (QOL).

DETAILED DESCRIPTION:
The purpose of this study is to clarify whether resecting pylorus-ring decreases delayed gastric emptying after pancreaticoduodenectomy and improves postoperative quality of life(QOL)compared with preserving pylorus-ring. Delayed gastric emptying after pancreaticoduodenectomy are important to affect the postoperative course and QOL. However, there is no report that demonstrates the postoperative course between resecting pylorus-ring and preserving pylorus-ring. We conducted a prospective randomized trial on 130 patients who underwent pancreaticoduodenectomy comparing resecting pylorus-ring and preserving pylorus-ring.

The primary endpoint was defined as the decrease of delayed gastric emptying. The secondary endpoints were QOL, mortality and morbidity, including pancreatic fistula, intra-abdominal hemorrhage, and intra-abdominal abscess. Patients were recruited into this study before surgery, on the basis of whether pancreatic head resection was anticipated at Wakayama Medical University Hospital(WMUH) for pancreatic head and periampullary disease, and appropriate informed consent was obtained. Exclusion criteria was 1) patients with severe complications which were possible to prolong hospital stay, 2) patients who were diagnosed inadequacy for this study by a physician, 3) patients with a previous gastric resection, and 4) patients without an informed consent.

ELIGIBILITY:
Inclusion Criteria:

* On the basis of whether pancreatic head resection was anticipated at WMUH for pancreatic head and periampullary disease, and appropriate informed consent was obtained.

Exclusion Criteria:

* Patients with severe complications which were possible to prolong hospital stay
* Patients who were diagnosed inadequacy for this study by a physician
* Patients who could not be placed a pancreatic stent tube
* Patients without an informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2005-10; Primary Completion 2009-05 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
delayed gastric empty after pancreaticoduodenectomy | 1 month

SECONDARY OUTCOMES:
evaluation of quality of life, early and late complications after pancreaticoduodenectomy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Manabu Kawai, MD, Study Director — Wakayama Medical University, School of Medicine, Second Department of Surgery
Locations (1):
- Second Department of Surgery, Wakayama Medical University, School of Medicine, 811-1 Kimiidera, Wakayama, Japan

REFERENCES:
- [Background] Tani M, Kawai M, Terasawa H, Ina S, Hirono S, Shimamoto T, Miyazawa M, Uchiyama K, Yamaue H. Prognostic factors for long-term survival in patients with locally invasive pancreatic cancer. J Hepatobiliary Pancreat Surg. 2007;14(6):545-50. doi: 10.1007/s00534-007-1209-6. Epub 2007 Nov 30. PMID 18040618
- [Background] Kawai M, Tani M, Ina S, Hirono S, Nishioka R, Miyazawa M, Uchiyama K, Shimamoto T, Yamaue H. CLIP method (preoperative CT image-assessed ligation of inferior pancreaticoduodenal artery) reduces intraoperative bleeding during pancreaticoduodenectomy. World J Surg. 2008 Jan;32(1):82-7. doi: 10.1007/s00268-007-9305-y. PMID 18027017
- [Background] Kawai M, Tani M, Terasawa H, Ina S, Hirono S, Nishioka R, Miyazawa M, Uchiyama K, Yamaue H. Early removal of prophylactic drains reduces the risk of intra-abdominal infections in patients with pancreatic head resection: prospective study for 104 consecutive patients. Ann Surg. 2006 Jul;244(1):1-7. doi: 10.1097/01.sla.0000218077.14035.a6. PMID 16794381
- [Background] Terasawa H, Uchiyama K, Tani M, Kawai M, Tsuji T, Tabuse K, Kobayashi Y, Taniguchi K, Yamaue H. Impact of lymph node metastasis on survival in patients with pathological T1 carcinoma of the ampulla of Vater. J Gastrointest Surg. 2006 Jun;10(6):823-8. doi: 10.1016/j.gassur.2006.01.013. PMID 16769538
- [Background] Tani M, Kawai M, Terasawa H, Ina S, Hirono S, Uchiyama K, Yamaue H. Does postoperative chemotherapy have a survival benefit for patients with pancreatic cancer? J Surg Oncol. 2006 May 1;93(6):485-90. doi: 10.1002/jso.20440. PMID 16615151
- [Background] Tani M, Terasawa H, Kawai M, Ina S, Hirono S, Uchiyama K, Yamaue H. Improvement of delayed gastric emptying in pylorus-preserving pancreaticoduodenectomy: results of a prospective, randomized, controlled trial. Ann Surg. 2006 Mar;243(3):316-20. doi: 10.1097/01.sla.0000201479.84934.ca. PMID 16495694
- [Background] Tani M, Kawai M, Terasawa H, Ueno M, Hama T, Hirono S, Ina S, Uchiyama K, Yamaue H. Complications with reconstruction procedures in pylorus-preserving pancreaticoduodenectomy. World J Surg. 2005 Jul;29(7):881-4. doi: 10.1007/s00268-005-7697-0. PMID 15951940
- [Background] Tani M, Onishi H, Kinoshita H, Kawai M, Ueno M, Hama T, Uchiyama K, Yamaue H. The evaluation of duct-to-mucosal pancreaticojejunostomy in pancreaticoduodenectomy. World J Surg. 2005 Jan;29(1):76-9. doi: 10.1007/s00268-004-7507-0. PMID 15592915
- [Background] Kawai M, Uchiyama K, Tani M, Onishi H, Kinoshita H, Ueno M, Hama T, Yamaue H. Clinicopathological features of malignant intraductal papillary mucinous tumors of the pancreas: the differential diagnosis from benign entities. Arch Surg. 2004 Feb;139(2):188-92. doi: 10.1001/archsurg.139.2.188. PMID 14769579
- [Background] Yamaue H, Tani M, Onishi H, Kinoshita H, Nakamori M, Yokoyama S, Iwahashi M, Uchiyama K. Locoregional chemotherapy for patients with pancreatic cancer intra-arterial adjuvant chemotherapy after pancreatectomy with portal vein resection. Pancreas. 2002 Nov;25(4):366-72. doi: 10.1097/00006676-200211000-00008. PMID 12409831
- [Derived] Kawai M, Tani M, Hirono S, Miyazawa M, Shimizu A, Uchiyama K, Yamaue H. Pylorus ring resection reduces delayed gastric emptying in patients undergoing pancreatoduodenectomy: a prospective, randomized, controlled trial of pylorus-resecting versus pylorus-preserving pancreatoduodenectomy. Ann Surg. 2011 Mar;253(3):495-501. doi: 10.1097/SLA.0b013e31820d98f1. PMID 21248633